CLINICAL TRIAL: NCT00105339
Title: Simplified Consent for HIV Vaccine Trials
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Sponsor
Other Study IDs: ATN 006
Record Dates: First submitted 2005-03-11; First posted 2005-03-14 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2016-02

CONDITIONS: Adolescent Behavior
Keywords: consent form, vaccine trial; Simplified consent form
MeSH Terms: conditions — Adolescent Behavior

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Illustration Style Preference Group: Ten participants at each site will be invited to attend a focus group to determine their comfort with and preference for one of four styles of illustration. The same two concepts will be presented in each of the four styles and ratings will be obtained from all participants. Detailed information on why participants rated each of the styles the way they did will also be obtained by reviewing comments on the rating sheets and audiotapes of the groups. Groups will be run by the study coordinator at the Florida and New York sites, and by Dannie Hoffman, protocol coordinator, in Los Angeles, using a focus group script developed by Dr. Murphy.
- Review of Draft Focus Group: Lori Perez will travel to each site from Westat and conduct Review of Draft Focus Groups with adolescents and young adults (n per site = approximately 10 - 15) to collect final feedback on the adolescent friendly version (present key pieces of the adolescent friendly version and obtain feedback on the wording and the illustrations). Based on the focus group feedback, the research team will finalize the adolescent friendly materials.
- Comprehension/Recall Assessment: The assessment will be read to the participants to preclude reading problems. Responses will be recorded by the interviewer on the assessment instrument.

SUMMARY:
The main goal of this project is to develop and evaluate a simplified version of an HIV vaccine trial consent form designed for high-risk adolescents. The process will include: (1) reducing reading grade level by simplifying sentence structure and decreasing the use of infrequently used words; (2) re-organizing and categorizing the material for improved flow; and (3) developing a set of pictures to emphasize key concepts in the material. These materials will be tested among small focus groups of high-risk adolescents. A pre-post test design will be used to compare the simplified, adolescent-tailored consent form to one currently used in the National Institute of Allergy and Infection Diseases (NIAID) Vaccine Trial Information Booklet.

DETAILED DESCRIPTION:
In the United States, there has already been widespread preparation for the HIV vaccine efficacy trials. Since the first HIV vaccine trial enrolled volunteers in 1988, there have been numerous clinical trials of different vaccine candidates studied through NIAID's vaccine evaluation program. Since the outcome of a prophylactic HIV vaccine trial depends in part on the compliance of volunteers, one major effort that has been made is to determine the readiness of several high-risk populations to participate in vaccine trials. Numerous studies on the feasibility and willingness to participate in an adult HIV vaccine trial have already been conducted.

Increased willingness to participate has been found to be associated with high-risk behaviors, lower education level, and being uninsured or covered by public insurance, as well as higher HIV incidence rates. Baseline knowledge of vaccine trial concepts was low among all of the populations studied.

One population for which a vaccine could be extremely efficacious is high-risk adolescents-- who face a lifetime of dealing with a chronic illness if infected with HIV. Adolescents at risk for HIV and therefore eligible and in need of a vaccine are likely to be low-income, poorly educated, and a disenfranchised population. Moreover, they are likely to have below-average reading and verbal comprehension skills, and difficulty with medical terminology. Issues of literacy and comprehension of informed consent become even more critical when dealing with populations with special vulnerabilities. To achieve truly informed consent for vaccine trials, Hodel (1994) has insisted that further research is crucial in determining what information is meaningful to potential participants in order for them to decide whether to participate. Potential HIV vaccine participants must fully understand complex concepts (e.g., that a person will test positive for HIV, even though they do not have the virus--they are "vaccine positive").

Children and adolescents have developmental limitations on their abilities to comprehend information. With some exceptions, the majority of IRBs require parental consent for research involving minors. Typically, parent or guardian permission for research on minors may not be solicited for research with substantially greater than minimal risk unless there is direct benefit to the minor with a risk-benefit ratio at least as good as available alternatives. There are also special considerations for involvement of adolescents in research where needs of parents and of the adolescents may conflict in terms of concerns about privacy.

Studies have suggested that simplifying the language and using short sentences have enhanced understanding. Other studies support the use of visual aids to enhance adolescent understanding and to enable adolescents to give truly informed consent.

The aims of the project are to randomize adolescents at risk for HIV to either a simplified adolescent-friendly prototype condition, or to the standard condition in order to determine:

1. if adolescents assigned to the simplified, adolescent-tailored prototype condition have significantly better comprehension scores than those assigned to the standard condition;
2. if adolescents assigned to the simplified, adolescent-tailored prototype condition have significantly better recall scores than those assigned to the standard condition;
3. if willingness to participate in a vaccine trial is significantly different among adolescents assigned to the simplified condition compared to the standard condition.

ELIGIBILITY:
Inclusion Criteria:

* Ages 15 to 19 years (self identified)
* At risk for HIV/AIDS as determined by responses to an anonymous screen for sexual risk
* Giving assent or consent, depending on age
* English-speaking

Exclusion Criteria:

* Non-English speaking
* Not shown to be at risk through use of screener
* Unwilling/unable to provide informed consent/assent

Ages: 15 Years to 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: A sample of high-risk adolescents from 3 ATU sites will be recruited for both sets of focus groups, the Illustration Style Preference Group (n = 30; 10 per site) and the Review of Draft Groups (n = 45; 15 per site), and for the Comprehension/Recall Trial (n = 180; 60 per site), for total of 255 participants.
Sampling Method: Non-Probability Sample
Enrollment: 255 (Actual)
Dates: Start 2003-12; Primary Completion 2004-02 (Actual); Study Completion 2004-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Debra Murphy, PhD, Study Chair — Adolescent Trials Network
Locations (3):
- United States (3):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Children's Diagnostic and Treatment Center, Fort Lauderdale, Florida
  - Mount Sinai Medical Center, New York, New York

REFERENCES:
- See also: ATN Website — http://www.atnonline.org